CLINICAL TRIAL: NCT05032508
Title: Efficacy of the Application of Xylocaine Impregnated Compress in Reducing Per-procedural Pain During Ultrasound-guided Infiltration of Trigger Finger: a Randomized, Double-blind Controlled Study (SAUTYLO)
Brief Title: Efficacy of the Application of Xylocaine Impregnated Compress in Reducing Per-procedural Pain During Ultrasound-guided Infiltration of Trigger Finger
Acronym: SAUTYLO
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Fondation de l'Avenir (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: APHP210094; 2021-002052-36 (EudraCT Number)
Record Dates: First submitted 2021-08-27; First posted 2021-09-02 (Actual); Last update posted 2022-11-08 (Actual); Status verified 2022-09

CONDITIONS: Trigger Finger
Keywords: Trigger Finger; Xylocaine
MeSH Terms: conditions — Trigger Finger Disorder

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- xylocaine (Experimental)
  Interventions: Drug: Lidocaïne Aguettant 20 mg/ml
- Placebo (Placebo Comparator)
  Interventions: Drug: NaCl 0,9%

INTERVENTIONS:
Drug: Lidocaïne Aguettant 20 mg/ml — Lidocaïne Aguettant 20 mg/ml, injectable solution, applied to the skin with an impregnated compress, applied 15 minutes before infiltration performed by an experienced operator.
  Arms: xylocaine
Drug: NaCl 0,9% — Placebo (NaCl 0,9%), applied to the skin with an impregnated compress, applied 15 minutes before infiltration performed by an experienced operator.
  Arms: Placebo

SUMMARY:
The purpose of this study is to assess the efficacy of Xylocaine impregnated compress in reducing per-procedural pain during ultrasound-guided infiltration of Trigger Finger

DETAILED DESCRIPTION:
Trigger finger ultrasound-guided infiltrations are frequent and painful invasive procedures.

However, there is no current recommendation for per-procedural pain management, and in the majority of cases, infiltration is performed without prior skin anesthesia.

Xylocaine patches are of controversial efficacy in pain acute management. In current practice, they are not prescribed in advance and they are not well adapted to the topography of the finger.

On the other hand, a recent study showed the interest of administering lidocaine 2% by J-tip, a needle-free injection technique not available in France, before infiltration of Trigger Finger.

The investigators hypothesize that an impregnated compress in Xylocaine 20 mg/ml injectable solution, applied 15 minutes before the procedure, would reduce per-procedural pain.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years or older
* Trigger Finger (clinically defined by painful difficulty or protrusion when extending the finger) with an ultrasound-guided infiltration of cortisone derivatives indication.
* Written consent
* Affiliation to a Social Security system
* Prior medical examination

Exclusion Criteria:

* Neurological conditions affecting the hand other than carpal tunnel syndrome
* Intra-articular infiltration of the hand or the wrist ≤ 2 months
* Allergy to Xylocaine
* Contraindication to Xylocaine or cortisone derivatives
* Cognitive or behavioral disorders that make assessment impossible
* Persons referred to in articles L 1121-5; 6; 8; 9 of the Public Health Code (protected adults, under guardianship or curatorship, etc)
* Pregnancy and breastfeeding; absence of contraceptive method for women of childbearing age
* Participant unable to speak, read and write French

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-06-07 (Actual); Primary Completion 2023-06-07 (Estimated); Study Completion 2023-06-07 (Estimated)

PRIMARY OUTCOMES:
Average pain intensity during the ultrasound-guided infiltration. | Day 0, immadiately after infiltration
  Evaluation assessed by self-administered pain numeric rating scale (0, no pain and 100, maximum pain).

SECONDARY OUTCOMES:
Adverse Events | Day 0
  Adverse events based on a self-administered open-ended question
Pain acceptance level in patients with trigger finger during the ultrasound-guided infiltration | Day 0
  Pain acceptance will be assessed according to the patient himself on a self-administered scale (0, not at all acceptable and 100, completely acceptable).
Pain acceptance level assessed by the operator during the ultrasound-guided infiltration of trigger finger | Day 0
  Pain acceptance will be assessed according to the operator, on a scale (0, not at all acceptable and 100, completely acceptable).

CONTACTS AND LOCATIONS:
Overall Officials: Henri GUERINI, MD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Cochin hospital, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided